CLINICAL TRIAL: NCT07035145
Title: A Registered Observational Cohort Study of Dysferlinopathy in China
Brief Title: Observational Cohort Study of Dysferlinopathy in China
Status: Completed | Type: Observational
Sponsor: Peking University First Hospital (Other)
Responsible Party: Principal Investigator, Meng YU, Dr., Peking University First Hospital
Other Study IDs: NSFC82301584
Record Dates: First submitted 2025-06-04; First posted 2025-06-24 (Actual); Last update posted 2025-06-24 (Actual); Status verified 2025-06

CONDITIONS: Dysferlinopathy
Keywords: phenotype; natural history; genotype
MeSH Terms: conditions — Dysferlinopathy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Biospecimen Retention: Samples With DNA — Serum, Plasma, DNA, and RNA.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Dysferlinopathy: All patients with dysferlinopathy in China, irrespective of age. These dysferlinopathy patients were diagnosed according to i) two (predicted) pathogenic variations in DYSF gene, ii) one (predicted) pathogenic variation plus either absent dysferlin protein expression on muscle immunoblot (muscle biopsy was performed at Peking University First Hospital).

SUMMARY:
The cohort data to be collected aims to evaluate the phenotype, disease progression, natural history, as well as molecular, genetic, and morphological characteristics of dysferlinopathies (LGMD2B/Miyoshi) in China, contributing to the development of clinical outcome measures and the identification of potential biomarkers for future clinical trials.

DETAILED DESCRIPTION:
Dysferlinopathy is an autosomal recessive myopathy caused by mutations in the DYSF gene. Dysferlinopathy represents a rare group of muscular dystrophies, characterized by the "core" phenotypes of Miyoshi Myopathy (MM), Limb-Girdle Muscular Dystrophy Type R2 (LGMDR2) and the rarer distal myopathy with anterior tibial involvement. As the disease progresses, involvement of both proximal and distal muscles is observed in many patients, deviating from the classic muscle weakness patterns of LGMD2B or Miyoshi Myopathy. In addition, the age at onset and the progression of muscle weakness exhibit considerable heterogeneity among patients. Compared to other types of muscular dystrophy, dysferlinopathy exhibits variable onset ages for wheelchair dependency and likely carries a lower risk of cardiac and respiratory complications. Therefore, detailed and regular assessments of motor function, along with follow-up, are essential for systematically understanding the disease progression and natural history of dysferlinopathy, as well as for providing data to support future clinical trials.

Dysferlinopathy is characterized by typical dystrophic pathological changes, including necrosis and regeneration of muscle fibers, hypertrophy and atrophy, as well as proliferation of connective tissue. The absence of DYSF protein expression on the sarcolemma is a key pathological hallmark and diagnostic criterion of dysferlinopathy. Moreover, inflammatory infiltration represents a significant pathological feature of this condition. Specific analysis of the immune environment in skeletal muscles may serve as a potential therapeutic target for dysferlinopathy in future research.

The Chinese dysferlinopathy patient registry is a nationwide, population-based observational cohort study encompassing dysferlinopathy patients across all age groups, collecting retrospective data at study entry and prospective data during follow-up. This registry is intended to contribute to the development of clinical outcome measures and the identification of potential biomarkers for future clinical trials.

ELIGIBILITY:
Inclusion Criteria:

* Male or female patients of all ages at baseline.
* Confirmed diagnosis of dysferlinopathy proven by i) two (predicted) pathogenic variations in DYSF gene, ii) one (predicted) pathogenic variation plus either absent dysferlin protein expression on muscle immunoblot. Mutations will be checked for pathogenicity via the UMD bioinformatics tools and and by checking the literature and mutation /variant databases.
* Ambulant with or without aids; or full-time wheelchair user, i.e. non-ambulant; with the ratio 2:1 between recruited ambulant and recruited non-ambulant patients.
* Ability to perform assessments (there will be different assessments for ambulant and non-ambulant patients).
* Informed consent to participate in the study.

Exclusion Criteria:

* Decline to participate.
* Other neuromuscular disease (such as Duchenne/Becker muscular dystrophy or Myotonic dystrophy).
* Serious systemic illness (such as cute cardiac, renal, hepatic insufficiency, myocardial infarction or an acute cerebrovascular accident (stroke) as well as infectious diseases).

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All patients with dysferlinopathy in China, irrespective of age. These dysferlinopathy patients were diagnosed according to i) two (predicted) pathogenic variations in DYSF gene, ii) one (predicted) pathogenic variation plus either absent dysferlin protein expression on muscle immunoblot (muscle biopsy was performed at Peking University First Hospital).
Sampling Method: Non-Probability Sample
Enrollment: 160 (Actual)
Dates: Start 2024-05-01 (Actual); Primary Completion 2025-03-15 (Actual); Study Completion 2025-03-31 (Actual)

PRIMARY OUTCOMES:
Clinical status of patients with dysferlinopathy (MMT score) | From date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 20 years
  Muscle strength will be assessed using MMT and will be expressed in points for each of the muscle groups assessed. Data will be reported from 0 to 5, with lower score pointing to weaker muscle strength.
North Star assessment for limb girdle-type muscular dystrophies (NSAD) in patients with dysferlinopathy | From date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 20 years
  A functional scale that will be used to measure motor performance in individuals with LGMD. Data will be reported from 0 to 54, with lower score pointing to worse motor performance.
Clinical status of patients with dysferlinopathy (6-minute walk test) | From date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 20 years
  The participant will be asked to complete maximal distance in 6 minute as quickly as safely possible and the time in seconds is recorded.

SECONDARY OUTCOMES:
Muscle MRI in patients with dysferlinopathy | At baseline and during patients visits and follow-up through study completion, an average of 1 year.
  To characterize muscle involvement based on MRI results; To evaluate the progression of muscle involvement based on repeated MRI during follow-up;
Muscle pathology analysis in patients with dysferlinopathy (dysferlin and inflammatory infiltration detection ) | Conducted with informed consent at baseline.
  Muscle biopsy samples were taken from the biceps brachii or quadriceps femoris. Serial frozen sections were stained with haematoxylin and eosin, modified Gomori trichrome, periodic acid-Schiff, oil red O, acid phosphatase enzyme, adenosine triphosphate enzyme (pH 4.5 and 10.8), nicotinamide adenine dinucleotide tetrazolium reductase, succinate dehydrogenase, and cytochrome c oxidase stains. The sections were immunohistochemically stained with primary antibodies against human dysferlin, desmin, major histocompatibility complex class-I, membrane attack complex (MAC), and CD cells (including CD3, CD4, CD8, CD20, and CD68).

CONTACTS AND LOCATIONS:
Locations (1):
- Peking University First Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided